CLINICAL TRIAL: NCT02596685
Title: Effects of Electronic Cigarette Use on the Human Lung
Brief Title: Effects of Electronic Cigarette Use on the Lungs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Peter Shields, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OSU-15098; NCI-2015-00842 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-10-08; First posted 2015-11-04 (Estimated); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Current Smoker; Never Smoker; Tobacco Use Disorder; Former Smoker; E-cig User
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Bronchoscopy; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (electronic-cigarette) (Experimental): Patients receive nicotine-free and flavor-free electronic cigarettes and instructed to use them BID over a 2 hour period for 4 weeks.
  Patients undergo a second bronchoscopy during week 5.
  Interventions: Procedure: Bronchoscopy; Other: Electronic Cigarette; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm B (control) (Experimental): Patients receive no intervention.
  Patients undergo a second bronchoscopy during week 5.
  Interventions: Procedure: Bronchoscopy; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm I (bronchoscopy of the left lung) (Experimental): Patients undergo bronchoscopy of the left lung over 30-60 minutes.
  Interventions: Procedure: Bronchoscopy; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm II (bronchoscopy of the right lung) (Experimental): Patients undergo bronchoscopy of the right lung over 30-60 minutes.
  Interventions: Procedure: Bronchoscopy; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Bronchoscopy — Undergo bronchoscopy
Other: Electronic Cigarette — Given nicotine-free and flavor-free electronic cigarettes
  Other Names: e-Cigarette; Electronic Nicotine Delivery System
  Arms: Arm A (electronic-cigarette)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies the effects of electronic cigarettes on the lungs. Studying the effects of electronic cigarettes on the lungs may provide the Food and Drug Administration (FDA) and other government regulators with important information, which may help in developing future regulations to make electronic cigarettes safer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1) To conduct a pilot cross-sectional study of e-cig users (n=16), never-smokers (n=8 - completed under an earlier version of the protocol before never-smokers were used for Aim 2), (newly added n=15), former smokers who have quit smoking and are currently not using e-cigs (n=15), former smokers who switched to e-cigs (n=15) and smokers (n=16) [total n=85), to better determine the influence of e-cig and smoking use (i.e., power) between never smokers and e-cig users, and to compare former smokers with e-cig use, and assessing use patterns and biomarkers by bronchoscopies using bronchioalveolar lavage (cell counts, inflammatory cytokines, untargeted metabolomics, and microbiome assessment), bronchial brushings (miRNA and mRNA expression, DNA methylation, acrolein DNA adducts, and mitochondrial DNA mutations and copy number variation), blood and urine to assess exposure to the e-cigs ingredients, saliva for oral microbiome assessment, and nasal brushing and nasal lavages for the lung toxicity as examined in this study as surrogate markers for the lung. We will also measure fractional exhaled nitric oxide (FeNO) as a marker of lower airway inflammation; and,

1a) Conduct a supplemental contamination study to measure if bacteria from oral cavity, nasal cavity or oropharynx may contaminate BAL fluid recovered during the bronchoscopy (n=30). Contamination analyses will measure if bacterial species found in oral cavity, nasal cavity and oropharynx are recovered in BAL. Contamination analyses will not examine differences between groups.

2) To conduct a 4 week pilot clinical trial of nicotine-free and flavor-free e-cig use in never-smokers (n=30), randomized to e-cig use (n=15) or control (no e-cig use) (n=15), and assess biomarkers as in Aim 1 by bronchoscopy at baseline and at 4 weeks while on product (week 5 of trial).

OUTLINE:

PART I: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo bronchoscopy of the left lung over 30-60 minutes.

ARM II: Patients undergo bronchoscopy of the right lung over 30-60 minutes.

PART II: Patients who are never-smokers are then randomized to 1 of 2 arms.

ARM A: Patients receive nicotine-free and flavor-free electronic cigarettes and instructed to use them twice daily (BID) over a 2 hour period for 4 weeks.

ARM B: Patients receive no intervention.

In both arms, patients undergo a second bronchoscopy during week 5.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1 only: 1) smokers who smoke at least 10 cigarettes per day with a stable smoking pattern of at least 6 months and no prior e-cig use within one year. Smoking status will be confirmed by salivary cotinine; subjects with at least 10 ng/ml cotinine in their saliva being considered smokers [150]. 2) e-cig users who report using e-cigs daily for 3 months with at least one nicotine-containing cartridge/day or 1 ml of liquid/day. They should have not smoked a cigarette for at least one year. 3) former smokers currently using nicotine-containing e-cigs who have completely switched to e-cigs 1-5 years earlier, and previously smoked >10 cigs/day for >1 year. 4) former-smokers who have quit smoking 1-5 years previously, and who previously smoked >10 cigs/day for >1 year and no e-cig use for a year and <10 days in their lifetime. 5) never-smokers who have smoked less than 100 cigarettes in their lifetime and not for at least 1 year, and not have used an e-cig for at least 1 year. Lack of regular smoking will be confirmed by NicAlert.
* Aim 2 only: Non-smokers who have smoked less than 100 cigarettes in their lifetime and not for at least 1 year, and not have used an e-cig for at least 1 year. Lack of regular smoking will be confirmed by salivary cotinine. Participants should be in good physical and mental health, particularly those randomized to the control condition;
* No unstable and significant medical conditions as determined by medical history (see exclusion criteria below) to ensure safety of the subject, to minimize the effects of poor health on biomarker measures and to maximize compliance to study procedures);
* Able to read adequately to complete the survey and related study documents or give consent; and
* Subject has provided written informed consent to participate in the study.

Exclusion Criteria:

* Immune system disorders, pulmonary diseases (e.g., asthma within the prior 5 years, acute bronchitis within 1 year, COPD, chronic bronchitis, and restrictive lung disease), clinically diagnosed kidney or liver diseases, or any other medical disorders that will increase the risk from bronchoscopy, affect biomarker data, or increase risk of an adverse effect from e-cig use. All subjects are screened by a pulmonologist obtaining a medical history and a physical examination (heart, lungs and oral cavity) to ensure no increased risk from bronchoscopy or e-cig use;
* General anesthesia within one year;
* Use of inhalant medications in the last 3 months;
* Use of antibiotics in prior 30 days;
* Use of steroids, including corticosteroids, in prior 30 days;
* Allergies to study medications, such as, lidocaine, Versed, Fentanyl or Cetacaine
* Bronchoscopy or any other lung procedure for any reason within the previous year;
* Current or recent (within three months) alcohol or drug abuse problems, including marijuana use within the last 30 days. Subjects with a positive Tetrahydrocannabinol (THC) strip test at any visit will be excluded;
* Other tobacco use (e.g., combustible products, vapors, etc.) within the last 3 months;
* Other tobacco use within the past year for 7 consecutive days or 14 times.
* Currently using nicotine replacement or other tobacco cessation products (to minimize confounding effects of another product) or intention to quit in next three months;
* BMI > 40 (risk of unstable airway)
* Pregnant or breastfeeding in prior 3 months - If the subject is female, the investigator will provide a urine pregnancy test at no cost to the subject. The subject will take the pregnancy test before each bronchoscopy; and,
* Unable to read for comprehension or completion of study documents.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Biomarker expression analysis to include cell counts | Up to week 5
  Using bronchoalveolar lavage, and bronchial brushings for gene expression use patterns and biomarkers will be assessed and compared between two groups (e.g., non-smokers vs. smokers). For univariable comparisons, non-parametric methods such as the Kruskal-Wallis H-test for more than two independent groups and the Mann Whitney U-test for two independent groups will be used. Group associations controlling for possible confounders or effect modifiers will be explored using multiple linear regression models.
Biomarker expression analysis to include inflammatory cytokines (Part I) | Up to week 5
  Using bronchoalveolar lavage, and bronchial brushings for gene expression use patterns and biomarkers will be assessed and compared between two groups (e.g., non-smokers vs. smokers). For univariable comparisons, non-parametric methods such as the Kruskal-Wallis H-test for more than two independent groups and the Mann Whitney U-test for two independent groups will be used. Group associations controlling for possible confounders or effect modifiers will be explored using multiple linear regression models.
Biomarker expression analysis to include untargeted metabolomics (Part I) | Up to week 5
  Using bronchoalveolar lavage, and bronchial brushings for gene expression use patterns and biomarkers will be assessed and compared between two groups (e.g., non-smokers vs. smokers). For univariable comparisons, non-parametric methods such as the Kruskal-Wallis H-test for more than two independent groups and the Mann Whitney U-test for two independent groups will be used. Group associations controlling for possible confounders or effect modifiers will be explored using multiple linear regression models.
Biomarker expression analysis to include gene expression (Part I) | Up to week 5
  Using bronchoalveolar lavage, and bronchial brushings for gene expression use patterns and biomarkers will be assessed and compared between two groups (e.g., non-smokers vs. smokers). For univariable comparisons, non-parametric methods such as the Kruskal-Wallis H-test for more than two independent groups and the Mann Whitney U-test for two independent groups will be used. Group associations controlling for possible confounders or effect modifiers will be explored using multiple linear regression models.
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment (Part II) | Baseline to 5 weeks
  Descriptive statistics and plots will be used to informally assess changes in biological parameters between bronchoscopies; repeated measures models may be used to control for possible confounding between the groups as well as provide estimates for future power calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Shields, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McElroy JP, Song MA, Barr JR, Gardner MS, Kinnebrew G, Kuklenyik Z, Kusovschi JD, Rees JC, Blount BC, Tsai M, Wewers MD, Kamel S, Reisinger SA, Singh A, Weng DY, Shields PG. Lung lipids associated with smoking and ECIG use in a cross-sectional study and clinical trial. Respir Res. 2025 May 20;26(1):193. doi: 10.1186/s12931-025-03267-w. PMID 40394619
- See also: The Jamesline — http://cancer.osu.edu